CLINICAL TRIAL: NCT00730470
Title: A Phase I, Open-label, Dose-Finding Study to Assess the Safety and Tolerability of U3-1287 (AMG 888), a Human Monoclonal Antibody Targeting HER3 in Patients With Advanced Solid Tumors.
Brief Title: Phase I Study of U3P1287/01, Including Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U3 Pharma GmbH (Industry)
Responsible Party: Dr Alan Boyd MD, U3 Pharma GmbH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U3P1287/01
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Advanced Solid Tumors
Keywords: Human Epidermal Growth Factor Receptor 3; HER3; Heregulin; erb B3; Solid Tumors; Phase I Clinical Study
MeSH Terms: conditions — Lethal Congenital Contracture Syndrome 2; Fibromatosis, Gingival, 2 | interventions — patritumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: U3-1287 (AMG888)

INTERVENTIONS:
Drug: U3-1287 (AMG888) — IV Infusion Dose Escalation (Part 1) - 5 Dose Cohorts Dose Expansion (Part 2) - 30 patients

SUMMARY:
This is a Phase 1 clinical study to investigate the safety, pharmacokinetics, and pharmacodynamics of U3-1287 (AMG 888), a fully human monoclonal antibody targeting the HER3 receptor, in patients with advanced solid tumors. Eligible patients will have disease that is refractory or resistant to standard treatments or for which no standard therapy exists. The study will be conducted in two parts; a dose escalation (Part 1) and a dose expansion (Part 2). The hypothesis for this study is that U3-1287 (AMG888) will be safe and well tolerated in patients with advanced solid tumors and will show initial evidence of anti-tumor activity.

ELIGIBILITY:
Key Inclusion Criteria:

* Pathologically or cytologically documented advanced solid tumor that is refractory to standard treatment, for which no standard therapy is available, or the patient refuses standard therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Men or women at least 18 years of age
* Adequate hematologic, cardiac, renal, hepatic, metabolic, and coagulation function

Key Exclusion Criteria:

* Presence of untreated or symptomatic brain metastasis.
* Presence of ascites or pleural effusion requiring chronic medical intervention.
* Uncontrolled hypertension
* Concurrent or previous (within 1 week of study day 1) anticoagulation therapy, except low-dose warfarin (≤ 2 mg/day) or low dose,low molecular weight heparin for prophylaxis against central venous catheter thrombosis.
* Recent major surgical procedure or not yet recovered from major surgery
* Recent participation in clinical drug trials.
* Participation in other investigational procedures.
* Unresolved toxicities from prior anti-cancer therapy
* Patient who is pregnant (e.g. positive human choriogonadotropin [HCG] test) or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of U3-1287 (AMG888) in patients with advanced solid tumors | Lenth of study
To evaluate maximum tolerated dose (MTD) of U3-1287(AMG888) when administered intravenously to patients with advanced solid tumors | Lenth of study

SECONDARY OUTCOMES:
Pharmacokinetic Parameters | Length of study
Pharmacodynamic Parameters | Length of study
Human anti-human antibody profile for U3-1287(AMG888) | Length of study

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Centre, New York, New York
  - Vanderbilt Ingram cancer Centre, Nashville, Tennessee
  - Northwest Medical Specialties, Tacoma, Washington

REFERENCES:
- [Derived] LoRusso P, Janne PA, Oliveira M, Rizvi N, Malburg L, Keedy V, Yee L, Copigneaux C, Hettmann T, Wu CY, Ang A, Halim AB, Beckman RA, Beaupre D, Berlin J. Phase I study of U3-1287, a fully human anti-HER3 monoclonal antibody, in patients with advanced solid tumors. Clin Cancer Res. 2013 Jun 1;19(11):3078-87. doi: 10.1158/1078-0432.CCR-12-3051. Epub 2013 Apr 16. PMID 23591447